CLINICAL TRIAL: NCT05919875
Title: Evaluating the Effectiveness of an Online 6-weeks Mindfulness-Based Cognitive Therapy in Depressed Sample: a Randomized Three-arm Clinical Trial
Brief Title: Online Mindfulness-Based Cognitive Therapy in Depressed Sample
Acronym: iMBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warsaw (Other)
Responsible Party: Principal Investigator, Jan Wardęszkiewicz, Msc, University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UWarsaw
Record Dates: First submitted 2023-05-31; First posted 2023-06-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2023-06

CONDITIONS: Moderate Depressive Episode; Mild Depressive Episode
Keywords: mindfulness-based cognitive therapy; depression; online intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Unguided iMBCT intervention (Experimental)
  Interventions: Behavioral: Unguided Mindfulness-Based Cognitive Therapy
- Guided iMBCT intervention (Experimental)
  Interventions: Behavioral: Guided Mindfulness-Based Cognitive Therapy
- Waiting list group (No Intervention)

INTERVENTIONS:
Behavioral: Unguided Mindfulness-Based Cognitive Therapy — The unguided iMBCT intervention is divided into six sessions. The sessions are an online adaptation of the regular MBCT. Subsequent sessions are unlocked gradually, once a week. The training consists of audio/video recordings and a workbook. Materials are recorded by a certified MBCT teacher and represent topics raised during regular courses:
  1. Awareness and automatic pilot
  2. Living in our heads
  3. Being present in the body
  4. Recognizing aversion
  5. Allowing / Letting be
  6. "How can I best take care of myself?"
  The intervention requires daily commitment of about 30-40 minutes.
  Arms: Unguided iMBCT intervention
Behavioral: Guided Mindfulness-Based Cognitive Therapy — The guided iMBCT intervention consists of six online meetings in groups of maximum 25 participants. The weekly meetings will be led by an experienced and certified MBCT teacher. The course of the meeting will represent thematically the unguided condition according to the agenda:
  * Introduction to the topic
  * Guided meditation
  * Brief inquiry and discussion
  * Setting tasks for the upcoming week
  To reduce the number of differences between the conditions as much as possible and narrow it down to the active participation of the teacher, the meetings will be modified version of MBCT and will last maximum 90 minutes. Between the meetings participants will be ask to practice daily 30-40 minutes mindfulness exercises.
  Arms: Guided iMBCT intervention

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the online 6-weeks Mindfulness-Based Cognitive Therapy (iMBCT) in depressed sample and compare the guided intervention to an unguided one. The main questions the study aims to answer are:

* To what extent completing iMBCT will reduce the severity of depressive symptoms in mild to moderately depressed sample?
* What are the differences in participants who completed the program or responded to treatment and those who discontinued it?
* What are the differences in treatment effect between two active conditions (guided and unguided iMBCT) and a passive one - waiting-list group?

Researchers will compare two iMBCT interventions with a waiting-list group to assess the therapeutic effects of iMBCT on depression, anxiety and other measures related to the mental health.

DETAILED DESCRIPTION:
Depression affects more than 300 millions of people worldwide and is perceived as a largest contributor to global disability (World Health Organisation, 2017). Although the research into depression has been expanding in the last decades (Ledford, 2014), the epidemiological data suggests that a prevalence trend is not decreasing (Ormel, Cuijpers, Jorm et al., 2020).

Standard treatment such as psychotherapy or pharmacotherapy is expensive and often associated with other barriers such as limited availability of specialists or waiting-lists (Biringer, Sundfør, Davidson, 2015), which stresses the importance of seeking and investigating other approaches that could address mentioned issues (Rudd & Beidas, 2020).

With the development of technology, online psychological interventions have been created to offer more accessible help. Among the various programs aimed at reduction of psychological distress, the ones based on cultivating mindfulness, are exponentially increasing in popularity (Lee, Kim, Webster et al., 2021).

One of the few most examined MBI's protocols, considered as "gold-standard" (Van Dam et al., 2018) is Mindfulness-Based Cognitive Therapy (MBCT, Teasdale, Segal, Williams, 2000). Recent meta-analysis has shown that the intervention could treat current episodes of depression (Goldberg, Tucker, Greene et al., 2019). In the latest National Institute for Clinical Excellence (2022) guidelines MBCT was listed as one of the first-choices for less severe depression.

Several studies demonstrated the effectiveness of the online version of MBCT (iMBCT) in treating depressive symptoms (Segal, Dimidjian, Boggs et al., 2020; Ritvo, Knyahnytska, Wang et al., 2021; Nissen, Zachariae, O'Connor et al., 2021), however the field is still fairly new and more research is needed to comprehensively evaluate the clinical utility of the intervention.

In this study the investigators decided to evaluate the effectiveness of two conditions of 6-weeks iMBCT (guided and unguided) and compare those two with a waiting-list group.

Individuals willing to take part in the study will complete an online screening test. Participants meeting the initical criterions - mild to moderate depressive symptoms - will be asked to take part in a structured clinical interview to increase the validity of the assessment and exclude those with comorbid psychiatric disorders.

Then after recruitment, participants will be randomized to one of the three mentioned above conditions. The unguided intervention will consist of the same thematic modules as guided one, however instead of online meetings materials will be uploaded on the platform.

Despite pre-test and post-test after six weeks, there will be follow-up measure after 3 months. Another outcome measure will be ecological momentary assessments taking place during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* meeting the screening criterions for depression
* confirmed diagnosis in the clinical interview - mild to moderate depressive episode
* 18 years old or older
* informed consent
* fluent in Polish
* willing to be randomized to intervention or waiting list group

Exclusion Criteria:

* lack of depressive symptoms constituting mild or moderate episode of depression
* suicidality
* severe depression
* current substance use disorder, psychotic disorders, bipolar
* current psychotherapy
* if antidepressant medication: has not been stable over the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Change in levels of depression - first tool | Baseline, week 6 and week 18
  The Patient Health Questionnaire (PHQ-9): It is a brief self-administered tool for screening and assessing depression severity according to the DSM criteria (Kroenke et al., 2001). Respondents rate the statements on a 4-points scale, yielding a score between 0 and 27.
Change in levels of depression - second tool | Baseline, week 6 and week 18
  To increase the reliability of diagnosis, second tool measuring depression will be used: The Center for Epidemiologic Studies Depression Scale (Radloff, 1977). It is a 20-item instrument with each item rated on a four-point scale ranging from 0 ("rarely or none of the time") to 3 ("most or all of the time").
Change in levels of anxiety | Baseline, week 6 and week 18
  Generalized Anxiety Disorder (GAD-7) scale: it is a brief tool that consists of seven items measuring worry and anxiety symptoms. (Spitzer et al., 2006). Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity.
Change in levels of self-compassion | Baseline, week 6 and week 18
  Self-compassion will be measured with a short form of Self-Compassion Scale (SCS-SF; Raes et al., 2011). The tool consists of 12 items (eg. 'I try to see my failings as part of the human condition.') to which person refers on a five-point scale.
Change in level of resilience | Baseline, week 6 and week 18
  The level of resilience will be computed with polish Resilience Measurement Scale (The Resiliency Assessment Scale, SPP-25; Ogińska - Bulik, Juczyński, 2008). The scale consists of 25 statements (e. g. I can easily adapt to new situations) to which respondent relates on a five-point Likert scale.
Change in levels of mindfulness | Baseline, week 6 and week 18
  Five Facet Mindfulness Questionnaire-15 (FFMQ-15): It is a short tool to measure mindfulness as a trait. The items will be measured on a 5-point Likert-type scale from 1 (never or rarely true) to 5 (very often or always true). Example items include: "I do jobs or tasks automatically without being aware of what I'm doing"

SECONDARY OUTCOMES:
Change in levels of rumination | Baseline, week 6 and week 18
  The Ruminative Response Scale (RRS): It is a 22-item tool measuring responses to depressed mood that are self-focused, symptom-focused, and focused on the possible causes and consequences of dysphoric mood (Nolen-Hoeksema & Morrow, 1991). Each item is rated on a Likert scale ranging from 1 (almost never) to 4 (almost always).
Change in levels of cognitive fusion | Baseline, week 6 and week 18
  The Cognitive Fusion Questionnaire (CFQ): It is a 7-item universal tool measuring cognitive fusion and was created as an alternative to questionnaires that were embedded in narrowed-down contexts, such as anxiety disorders or youth (Gillanders et al., 2014).
Change in levels of experiential avoidance | Baseline, week 6 and week 18
  The Brief Experiential Avoidance Questionnaire (BEAQ): It is a 15-items assessment that was created to measure EA (Gámez et al., 2014). Participants respond to the statements on a 6-point Likert scale (1: "strongly disagree"; 6: "strongly agree").

OTHER OUTCOMES:
Ecological momentary assessment | Week 1,2 and 6
  EMA is a process measure that allows to deepen the understanding of mechanisms of change in the intervention. Our EMA consists of:
  * 4 questions about depression
  * 3 questions about mindfulness
  * 4 questions about ruminations
  * 1 affect scale
Working Alliance | week 2
  Working Alliance Inventory tailored to the Internet condition (WAI-TECH-SF): it is a 12-item questionnaire designed to assess the therapeutic alliance with the online program. Participants will response on a seven-point Likert scale, ranging from 1 (never) to 7 (always) (Herrero at al., 2020).
Credibility and Expectancy | week 2
  Credibility and Expectancy Questionnaire (CEQ) is a 6-item tool assessing treatment expectancy based on the participant's beliefs. The questionnaire consists of two factors: expectancy (with three questions rated on a 10-point scale, ranging from 1 to 9) and credibility (with one question rated on a 10-point scale and two questions rated on a 1-100% scale) (Devilly, Borkovec, 2000).
Attitudes towards Psychological Online Interventions | Baseline
  The Attitudes towards Psychological Online Interventions Questionnaire (APOI): it is a 16-item tool that was created to assesses respondents' acceptance of Internet interventions along four dimensions (Skepticism and Perception of Risks, Confidence in Effectiveness, Technologization Threat, and Anonymity Benefits). The answers are collected on a five-point Likert-scale (1 = totally agree, 2 = rather agree, 3 = not sure, 4 = rather disagree, 5 = totally disagree)(Schröder et al. 2015) .
Locus of Control in Well-Being | Baseline
  A Locus of Control Specific to Well-Being (WB-LOC12): it is a 12-item tool that aims to identify the patients' beliefs concerning the main forces influencing their well-being (Farnier et al., 2021)
Social support | Baseline
  The Multidimensional Scale of Perceived Social Support (MSPSS:it is a 12-item tool developed by Zimet and collaborators (1988) as a self-report measure to assess per- ceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Wardęszkiewicz, MSc, Principal Investigator — University of Warsaw; Paweł Holas, Ph.D., Study Chair — University of Warsaw
Locations (1):
- University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
We will provide data upon reasonable request.

REFERENCES:
- [Background] Surewicz WK. Effect of osmotic gradient on the physical properties of membrane lipids in liposomes. Chem Phys Lipids. 1983 Jul;33(1):81-5. doi: 10.1016/0009-3084(83)90010-5. PMID 6313244
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Wampold BE, Kearney DJ, Simpson TL. Mindfulness-based interventions for psychiatric disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2018 Feb;59:52-60. doi: 10.1016/j.cpr.2017.10.011. Epub 2017 Nov 8. PMID 29126747
- [Background] Segal ZV, Dimidjian S, Beck A, Boggs JM, Vanderkruik R, Metcalf CA, Gallop R, Felder JN, Levy J. Outcomes of Online Mindfulness-Based Cognitive Therapy for Patients With Residual Depressive Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Jun 1;77(6):563-573. doi: 10.1001/jamapsychiatry.2019.4693. PMID 31995132
- [Background] Chariyalertsak S, Sugano K, Ohkura H, Mori Y. Comparison of c-erbB-2 oncoprotein expression in tissue and serum of patients with stomach cancer. Tumour Biol. 1994;15(5):294-303. doi: 10.1159/000217904. PMID 7991990